CLINICAL TRIAL: NCT00006054
Title: Allogeneic Bone Marrow Transplantation in Patients With Primary Immunodeficiencies
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Fairview University Medical Center (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/15104; UMN-MT-1995-26; UMN-MT-9526
Record Dates: First submitted 2000-07-05; First posted 2000-07-06 (Estimated); Last update posted 2009-10-15 (Estimated); Status verified 2003-10

CONDITIONS: Immunologic Deficiency Syndromes; Chediak-Higashi Syndrome; Common Variable Immunodeficiency; Graft Versus Host Disease; X-Linked Lymphoproliferative Syndrome; Familial Erythrophagocytic Lymphohistiocytosis; Hemophagocytic Lymphohistiocytosis; X-linked Agammaglobulinemia; Wiskott-Aldrich Syndrome; Chronic Granulomatous Disease; X-linked Hyper IgM Syndrome; Severe Combined Immunodeficiency; Leukocyte Adhesion Deficiency Syndrome; Virus-Associated Hemophagocytic Syndrome
Keywords: Chediak-Higashi syndrome; Langerhans cell histiocytosis; Wiskott-Aldrich syndrome; X-linked agammaglobulinemia; X-linked hyper IgM syndrome; X-linked lymphoproliferative syndrome; chronic granulomatous disease; common variable immunodeficiency; complement deficiency; disease-related problem/condition; familial erythrophagocytic lymphohistiocytosis; genetic diseases and dysmorphic syndromes; graft versus host disease; hematologic disorders; hemophagocytic lymphohistiocytosis; histiocytosis; immunologic disorders and infectious disorders; leukocyte adhesion deficiency syndrome; primary immunodeficiency disease; rare disease; severe combined immunodeficiency; virus-associated hemophagocytic syndrome
MeSH Terms: conditions — Immunologic Deficiency Syndromes; Chediak-Higashi Syndrome; Common Variable Immunodeficiency; Graft vs Host Disease; Lymphoproliferative Disorders; Lymphohistiocytosis, Hemophagocytic; Bruton type agammaglobulinemia; Wiskott-Aldrich Syndrome; Granulomatous Disease, Chronic; Hyper-IgM Immunodeficiency Syndrome, Type 1; Severe Combined Immunodeficiency; Leukocyte-Adhesion Deficiency Syndrome; Histiocytosis, Langerhans-Cell; Hereditary Complement Deficiency Diseases; Genetic Diseases, Inborn; Hematologic Diseases; Histiocytosis; Immune System Diseases; Communicable Diseases; Primary Immunodeficiency Diseases; Rare Diseases | interventions — Antilymphocyte Serum; Busulfan; Cyclophosphamide; Cyclosporine; Etoposide; Methotrexate; Methylprednisolone; Prednisone

INTERVENTIONS:
Drug: anti-thymocyte globulin
Drug: busulfan
Drug: cyclophosphamide
Drug: cyclosporine
Drug: etoposide
Drug: methotrexate
Drug: methylprednisolone
Drug: prednisone
Procedure: Allogeneic Bone Marrow Transplantation

SUMMARY:
OBJECTIVES: I. Provide curative immunoreconstituting allogeneic bone marrow transplantation for patients with primary immunodeficiencies.

II. Determine relevant outcomes of this treatment in these patients including quality of survival, extent of morbidity and mortality from complications of the treatment (e.g., graft versus host disease, regimen related toxicities, B- cell lymphoproliferative disease), and completeness of functional immunoreconstitution.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients with severe combined immunodeficiency (SCID) using a matched sibling donor receive allogeneic bone marrow or umbilical cord blood transplantation on day 0. Patients receive graft versus host disease (GVHD) prophylaxis with methotrexate IV on days 1, 3, 6, and 11 and cyclosporine IV on days -3 to 50.

Patients with SCID using donors other than histocompatible siblings, Wiskott Aldrich syndrome using a histocompatible sibling donor, Wiskott Aldrich syndrome and under 5 years of age using donors other than histocompatible siblings, X-linked CD40 ligand deficiency using a histocompatible sibling donor, X-linked CD40 ligand deficiency and under 5 years of age using donors other than histocompatible siblings, other primary immunodeficiencies without manifestations of hemophagocytosis using a histocompatible sibling donor, or other primary immunodeficiencies without manifestations of hemophagocytosis and under 5 years of age using donors other than histocompatible siblings receive busulfan IV over 2 hours every 6 hours on days -9 to -6, cyclophosphamide IV on days -5 to -2, and antithymocyte globulin (ATG) twice daily on days -4 to -1. Allogeneic bone marrow or umbilical cord blood transplantation takes place on day 0. Patients receive graft versus host disease (GVHD) prophylaxis with methotrexate IV on days 1, 3, 6, and 11 and cyclosporine IV on days -3 to 50.

Patients with hemophagocytic lymphohistiocytosis, Chediak Higashi syndrome, X-linked lymphoproliferative syndrome, severe progressive Langerhans cell histiocytosis, or other primary immunodeficiencies with complications of hemophagocytosis receive busulfan IV over 2 hours every 6 hours on days -9 to -6, cyclophosphamide IV over 2 hours on days -5 to -2, etoposide IV over 22 hours on days -5 to -3, and ATG IV twice daily on days -2, -1, 1, and 2. Allogeneic bone marrow or umbilical cord blood transplantation takes place on day 0. Patients receive graft versus host disease (GVHD) prophylaxis with methotrexate IV on days 1, 3, 6, and 11 and cyclosporine IV on days -3 to 50.

Patients with Wiskott Aldrich syndrome or other primary immunodeficiencies without manifestations of hemophagocytosis, who are over 5 years of age and using donors other than histocompatible siblings, receive busulfan IV over 2 hours every 6 hours on days -6 and -5, cyclophosphamide IV over 2 hours on days -4 and -3, total body irradiation on day -2, and ATG IV over 2 hours twice daily on days -2, -1, 2, and 3. Allogeneic bone marrow or umbilical cord blood transplantation takes place on days 0 and 1. Patients receive GVHD prophylaxis with methylprednisolone IV every 12 hours on days 2-21, oral prednisone every 12 hours on days 22-100 and then tapered off over days 101 to 128, and cyclosporine IV over 2 hours every 8-12 hours on days -3 to 100.

All patients are followed as determined by their primary physician.

ELIGIBILITY:
* Severe combined immunodeficiency All ages with histocompatible sibling donors or with other donors OR Wiskott Aldrich syndrome All ages with histocompatible sibling donors or with other donors OR X-linked CD40 ligand deficiency All ages with histocompatible sibling donors OR Under 5 years of age with donors other than histocompatible siblings OR Other primary immunodeficiencies without manifestations of hemophagocytosis All ages with histocompatible sibling donors or with other donors OR Hemophagocytic lymphohistiocytosis (HLH) Familial erythrophagocytic lymphohistiocytosis (FEL), familial HLH (FHLH), recurrent virus-associated hemophagocytic syndrome (VAHS) All ages with related or unrelated donors OR Chediak Higashi syndrome All ages with related or unrelated donors OR X-linked lymphoproliferative syndrome All ages with related or unrelated donors OR Other primary immunodeficiencies with complication of hemophagocytosis All ages with related or unrelated donors OR Severe progressive Langerhans cell histiocytosis All ages with related or unrelated donors

Max Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 2000-03; Primary Completion 2002-12 (Actual); Study Completion 2002-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: K. Scott Baker, Study Chair — Fairview University Medical Center
Locations (1):
- Fairview University Medical Center, Minneapolis, Minnesota, United States